CLINICAL TRIAL: NCT00012740
Title: A Casefinding and Referral System for Older Veterans Within Primary Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IIR 95-050
Record Dates: First submitted 2001-03-14; First posted 2001-03-16 (Estimated); Last update posted 2015-04-07 (Estimated); Status verified 2005-12

CONDITIONS: Depression; Incontinence; Cognitive Impairment
MeSH Terms: conditions — Depression; Cognitive Dysfunction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Arm 1 (Other)
  Interventions: Behavioral: Casefinding and Referral System

INTERVENTIONS:
Behavioral: Casefinding and Referral System

SUMMARY:
Underdiagnosis and undertreatment of elderly persons remains a widespread problem. While many innovative geriatric care programs exist within VHA, we still lack a systematic process for identifying at-risk elders from the larger VA population who are likely to benefit from specialized geriatric services.

DETAILED DESCRIPTION:
Background:

Underdiagnosis and undertreatment of elderly persons remains a widespread problem. While many innovative geriatric care programs exist within VHA, we still lack a systematic process for identifying at-risk elders from the larger VA population who are likely to benefit from specialized geriatric services.

Objectives:

Our goal is to improve care for at-risk older veterans through a comprehensive system of casefinding, assessment, referral and follow-up within the primary care setting. We hypothesize that subjects receiving this intervention will have more complete evaluation and treatment for selected geriatric conditions (i.e., falls, urinary incontinence, functional status impairments, depression, and cognitive deficits), better continuity of care, less decline in functional status, and better general health than subjects receiving usual care.

Methods:

This randomized controlled trial is being performed at the Sepulveda VA Outpatient Clinic. The study sample is composed of community-dwelling veterans aged 65 and older who are not receiving VA geriatric services. Veterans are mailed a health screening survey to identify those at risk for decline based on criteria established in pilot work. At-risk respondents who are in the intervention group receive a structured telephone assessment (casefinding) and referral to appropriate geriatric services, including a geriatric assessment and teaching clinic integrated with primary care, and telephone case management. Subjects in the control group receive usual care. Major outcome measures collected by telephone interview at baseline, 12, 24, and 36 months include functional status, self-rated health, satisfaction, and health care utilization. Medical records are reviewed for evidence of evaluation and treatment of the target conditions.

Status:

Data collection for this project was completed on September 30, 2001. The subject recruitment phase was completed in August, 1998. Collection of 36 month follow-up data has been completed for all subjects enrolled. Data analysis and preparation of publication is in press.

ELIGIBILITY:
Inclusion Criteria:

Subjects have to have a score of 4 or higher in a screening questionnaire and have been seen at clinic in the past 18 months.

Exclusion Criteria:

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 792 (Estimated)
Dates: Study Completion 2001-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Laurence Z. Rubenstein, MD MPH, Principal Investigator — VA Greater Los Angeles Healthcare System, Sepulveda, CA; Cathy A. Alessi, MD, Principal Investigator — VA Greater Los Angeles Healthcare System, Sepulveda, CA
Locations (1):
- VA Greater Los Angeles Healthcare System, Sepulveda, CA, Sepulveda, California, United States

REFERENCES:
- [Result] Alessi CA, Josephson KR, Harker JO, Pietruszka FM, Hoyl MT, Rubenstein LZ. The yield, reliability, and validity of a postal survey for screening community-dwelling older people. J Am Geriatr Soc. 2003 Feb;51(2):194-202. doi: 10.1046/j.1532-5415.2003.51058.x. PMID 12558716
- [Result] Hoyl MT, Alessi CA, Harker JO, Josephson KR, Pietruszka FM, Koelfgen M, Mervis JR, Fitten LJ, Rubenstein LZ. Development and testing of a five-item version of the Geriatric Depression Scale. J Am Geriatr Soc. 1999 Jul;47(7):873-8. doi: 10.1111/j.1532-5415.1999.tb03848.x. PMID 10404935